CLINICAL TRIAL: NCT05920174
Title: A Prospective Clinical Trial to Evaluate the Safety and Efficacy of an Implantable Neural Acquisitor & Stimulator System in Patients With Motor Disability
Brief Title: Clinical Trial to Evaluate the Safety and Efficacy of an Implantable Neural Acquisitor & Stimulator System in Patients With Motor Disability
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuracle Medical Technology(Shanghai) Co.,Ltd. (Industry)
Collaborators: Xuanwu Hospital, Beijing (Other); Beijing Tiantan Hospital (Other); Chinese PLA General Hospital (Other); Huashan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FABRK202301
Record Dates: First submitted 2023-05-29; First posted 2023-06-27 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Tetraplegia
MeSH Terms: conditions — Quadriplegia

STUDY DESIGN:
Intervention Model Description: an implantable neural acquisitor & stimulator system
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single (Experimental): Patients with motor disability（Complete or incomplete quadriplegia due to spinal cord injury, brain stem stroke, amyotrophic lateral sclerosis and other motor neuron disorders).
  Implantation of NEO device.
  Interventions: Device: NEO

INTERVENTIONS:
Device: NEO — Subjects will be implanted with the NEO device.

SUMMARY:
Through brain-computer interface alternative technology, patients can control the external equipment（wheelchairs, robotic arms, the WeChat app and other physical aids）with brain signals to improve the patients quality of life.

DETAILED DESCRIPTION:
To evaluate the safety and efficacy of an implantable neural acquisitor & stimulator system in patients with motor disability（Complete or incomplete quadriplegia due to spinal cord injury, brain stem stroke, amyotrophic lateral sclerosis and other motor neuron disorders).

Through brain-computer interface alternative technology, patients can control the external equipment（wheelchairs, robotic arms, the WeChat app and other physical aids）with brain signals to improve the patients quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 80 years of age;
2. Complete or incomplete quadriplegia due to spinal cord injury, brain stem stroke, amyotrophic lateral sclerosis and other motor neuron disorders;
3. After the neurological assessment, the brain motor-related cortex is functional, and there is no obvious organic disease or functional disease；
4. The above diseases have been diagnosed for at least 12 months and stable for at least 6 months after standard treatment；
5. The patient had normal cognitive function, good compliance and volunteered to participate in the clinical trial.

Exclusion Criteria:

1. Visual impairment such that extended viewing of a computer monitor would be difficult even with ordinary corrective lenses；
2. Combined with progressive neurological disease；
3. Combined with surgical contraindications identified by surgeons and anesthesiologists;
4. Participating in other clinical trials;
5. Other conditions deemed inappropriate by investigators and medical staff.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 12 months after implantation
  Number of Participants With the device-Related Adverse Events

SECONDARY OUTCOMES:
BCI performance classification accuracy | 3, 6, 12 months after implantation
  Achieved performance on BCI at conclusion of BCI sessions for each subject. Measured by classification accuracy (percentage of patient correct commands to overall number of detected commands)
BCI performance by bit rate | 3, 6, 12 months after implantation
  Achieved performance on BCI at conclusion of BCI sessions for each subject. Measured by bit rate (number of commands per minute).
Hours use of the implantable neural acquisitor & stimulator (NEO) per month | 3, 6, 12 months after implantation
  Hours use of the implantable neural acquisitor & stimulator (NEO) per month
Patient/caregiver satisfaction | 3, 6, 12 months after implantation
  The evaluation of patient and caregiver satisfaction will be carried out using a "satisfaction questionnaire" designed by the researcher (rated from Level 1 to 5) on their feelings (patient/caregiver) of use.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital，Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No